CLINICAL TRIAL: NCT05265169
Title: Ablation With Confirmation of Colorectal Liver Metastases (ACCLAIM) Prospective Trial for Microwave Ablation as a Local Cure
Brief Title: Ablation With Confirmation of Colorectal Liver Metastases (ACCLAIM)
Acronym: ACCLAIM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Society of Interventional Oncology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SIO-2021-01
Record Dates: First submitted 2022-02-22; First posted 2022-03-03 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Colorectal Liver Metastases

STUDY DESIGN:
Intervention Model Description: Prospective, open-label multicenter trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Microwave ablation with margin confirmation (Experimental): Patients who meet the eligibility criteria will undergo microwave ablation (MWA) of 1-3 colorectal cancer metastases with any FDA cleared/CE Marked Microwave Ablation System in accordance with the study site's standard-of-care (SOC) practices.
  Interventions: Device: Microwave ablation

INTERVENTIONS:
Device: Microwave ablation — Microwave ablation of colorectal liver metastases (CLM)

SUMMARY:
To demonstrate that microwave ablation (MWA) of up to 3 hepatic metastases, each with a maximum diameter of ≤ 2.5 cm will result in a 2-year local progression free survival of at least 90%. This is a standard of care (SOC) study.

DETAILED DESCRIPTION:
In this prospective, multi-center, standard of care trial we propose to establish microwave ablation (MWA) as the preferred curative therapy for selected colorectal liver metastases (CLM) that can be ablated with sufficient margins. Our hypothesis is that MWA of CLM ≤ 2.5 cm with confirmation of ablation margin over 5 mm achieves definitive local tumor control (local cure) with minimal morbidity.

This international study will enroll subjects with one to three CLMs (for a total of 330 tumors/approximately 275 subjects) eligible for local cure using MWA. Any FDA cleared or CE Marked MWA device will be acceptable for use. MWA will be performed with the intent to create a minimum margin of ablation of 5.0 mm and ideally ≥10 mm from the edge of the target tumor to the ablation periphery.

Minimum margin (MM) size will be documented intra-procedurally (immediately post MWA with contrast-enhanced CT) and again within 4-8 weeks after MWA. Assessment of the MM will be conducted by an independent core lab using an FDA approved/cleared image-processing software to provide 3D assessment of the ablation zone and margin.

* The initial assessment of the MM by the core lab will be conducted within 7 days of the MWA and again within 7 days after SOC imaging 4-8 weeks post MWA
* A minimal ablation margin of 5.0 mm will represent the necessary condition for technical success of the ablation.
* Margin assessment will be verified by an independent physician reviewer. For MMs less than 5 mm, repeat MWA will be performed whenever feasible/safe, within 30 days from detection, in order to achieve sufficient MM (> 5mm). Minimum margin size will be correlated with time to local tumor progression. Local disease-free progression (within or abutting the ablation zone) and hepatic disease-free survival (accounting for all tumors ablated) stratified by MM of ≥ 5.0-9.9 mm and ≥ 10.0 mm will be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must be at least 18 years old.
2. Patient has signed a written informed consent for the MWA and participation in the study.
3. Patient with pathologically confirmed CRC with hepatic metastases confirmed on imaging (e.g., CT or MRI).
4. Patient has up to 3 hepatic metastases, each up to 2.5 cm in largest diameter.
5. Patient may have up to 5 lesions in the lung (none larger than ≥ 2.0 cm) and/or any lymph node ≤2.0 cm in the largest diameter
6. Ability to safely create an ablation zone (AZ) that completely covers the tumor with minimal margin of 5.0 mm. Subcapsular (any tumor within 10 mm from the liver capsule) or perivascular (any tumor within 10 mm from a vessel larger than 3 mm) lesions may be included. For these tumors, the calculation of the margin will not apply to the area abutting the capsule or the vessel.
7. The target tumor(s) is/are visible by US and/or CT in a location where MWA is technically achievable and safe based on the proximity to adjacent structures. Protective maneuvers such as hydrodissection for organ mobilization are allowed and will be recorded.
8. ECOG performance status of 0-1.
9. Platelet count >50,000/mm3 (correctable allowed) within 30 days prior to study treatment.

Exclusion Criteria:

1. Patient is unable to lie flat or has respiratory distress at rest.
2. Patient has uncontrolled and uncorrectable coagulopathy or bleeding disorders.
3. Patient has a history of an allergic reaction to intravenous iodine that cannot be pre-medicated or prevents performance of a CT with IV contrast.
4. Patient has evidence of active systemic infection.
5. Patient has a debilitating medical or psychiatric illness that would preclude giving informed consent or receiving optimal treatment or follow up.
6. Patient is currently participating in other experimental studies that could affect the primary endpoint.
7. Patient unable to receive general anesthesia or adequate analgesia and sedation.
8. Tumor location less than 25 mm from hilum (see diagrams with illustration of central ducts).
9. Patient is currently pregnant or intends to become pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 275 (Estimated)
Dates: Start 2023-01-13 (Actual); Primary Completion 2027-11-11 (Estimated); Study Completion 2027-12-10 (Estimated)

PRIMARY OUTCOMES:
Local tumor progression free survival at 24 months | 24 Months
  See Above

SECONDARY OUTCOMES:
Hepatic progression free survival by Kaplan-Meier estimate | 24 Months
  See Above
Local tumor progression free survival between sufficient (5.0-9.9 mm) and ideal (≥10 mm) ablation margin categories using Kaplan-Meier methodology and the log-rank test | 24 Months
  See Above
Progression free survival using Kaplan-Meier methodology and the log-rank test | 24 Months
  See Above
Overall and disease specific survival following MWA using Kaplan-Meier methodology | 24 Months
  See Above
Proportion of target tumors treated with an ablation zone (AZ) that completely covers the target tumor(s) with minimal margin (MM) of at least 5 mm | 24 Months
  See Above
Proportion of subjects with CTCAE grade 3 events or greater within 90 days after MWA | 90 Days
  See Above

CONTACTS AND LOCATIONS:
Overall Officials: Constantinos Sofocleous, MD, PhD, FSIR, FCIRSE, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (5):
  - Miami Cancer Institute, Miami, Florida
  - Mayo Clinic, Rochester, Minnesota
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - MD Anderson Cancer Center, Houston, Texas
  - Medical College of WI, Milwaukee, Wisconsin
- National and Kapodistrian University of Athens (NKUA), Athens, Greece
- Amsterdam UMC, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sofocleous CT, Callstrom MR, Petre EN, Gonen M, Rilling WS, Ahmed M, Kelekis A, Soulen MC, Pereira P, Crocetti L, Dupuy DE, Solbiati L. Real-time 3D confirmation of complete ablation with margins as a local cure for colorectal liver metastases: the ACCLAIM trial. Trials. 2025 Sep 26;26(1):360. doi: 10.1186/s13063-025-09006-2. PMID 41013745